CLINICAL TRIAL: NCT03898063
Title: An Experimental Investigation of the Effects of an Entertainment Education Short Film on Internalized HIV-related Stigma, Sexual Partner Status Disclosure, and Medical Adherence Intentions Among Black HIV-positive Women in Miami-Dade County
Brief Title: 90 DAYS: An Entertainment Education Intervention to Evaluate a Short Film About HIV Status Disclosure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nicholas Carcioppolo, Assistant Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20170967; CTSI-Pilot-FY19-01 (Other Grant/Funding Number: University of Miami CTSI)
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): participants will receive a standard-of-care brochure detailing HIV status disclosure.
  Interventions: Behavioral: HIV pamphlet on disclosure
- intervention: 90 DAYS film (Experimental): participants will watch the film, 90 DAYS
  Interventions: Behavioral: 90 DAYS film

INTERVENTIONS:
Behavioral: 90 DAYS film — the intervention conditions include exposure to a film, 90 DAYS (approx 20 minutes long), an entertainment film detailing a woman's decision to tell her romantic partner that she is HIV-positive.
  Arms: intervention: 90 DAYS film
Behavioral: HIV pamphlet on disclosure — A standard-of-care brochure given to newly diagnosed HIV patients about the importance of status disclosure
  Arms: Control

SUMMARY:
This investigation seeks to understand if and how, the 90 Days film can be used as an intervention to address HIV-related stigmas, intimate partner status disclosure and HIV ART medical adherence among Black HIV positive women.

ELIGIBILITY:
Inclusion Criteria:

* Black women ages 18-50
* clinically diagnosed with HIV/AIDS
* Speak and comprehend English

Exclusion Criteria:

* pregnant women

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Carcioppolo, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Medical Campus, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention: 90 DAYS Film
Started | 74 | 74
Completed | 64 | 66
Not Completed | 10 | 8
Not completed — Withdrawal by Subject | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention: 90 DAYS Film | Total
Number analyzed (Participants) | 74 | 74 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.64 (6.65) | 32.64 (7.73) | 32.15 (7.21)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  sex: female | 64 | 66 | 130
  sex: male | 0 | 0 | 0
  sex: not reported | 10 | 8 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 74 | 74 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 64 | 66 | 130
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: HIV Self-stigmatization as Assessed Via Self Stigmatization Questionnaire
Description: self-report measure of the extent to which participants stigmatize themselves for being HIV positive. Quantified in the manuscript using the mean of the self-report scale. Scores range from 1-5 with higher scores indicating higher perceptions of self-stigmatization.
Time Frame: Day 1 post test
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: The participants in the control arm reviewed a brochure. After completing the pre-test, the randomize feature in Qualtrics, randomly assigned participants to one of two arms: control (brochure) or treatment (90 DAYS narrative).
- Treatment: The participants in the treatment arm viewed the 90 DAYS entertainment education film. After completing the pre-test, the randomize feature in Qualtrics, randomly assigned participants to one of two study arms: control (brochure) or treatment (90 DAYS film).
Arm/Group | Control | Treatment
Number analyzed (Participants) | 64 | 66
score on a scale | 2.93 (1.07) | 2.95 (1.14)

2. Primary Outcome: HIV Disclosure Intentions as Assessed by Disclosure Intentions Scale
Description: Self-report measure of the extent to which participants intend to disclose their HIV status to a partner. Quantified in the manuscript using the mean of the self-report scale. Scores range from 1-5 with higher scores indicating higher intentions of status disclosure.
Time Frame: Day 1 post-test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 64 | 66
score on a scale | 4.19 (0.82) | 4.45 (0.66)

3. Primary Outcome: Medical Adherence Intentions as Measured by the Medical Adherence Scale
Description: Self-report measure of participants likeliness to miss doses of their antiretroviral medication over a 30 day period. Quantified in the manuscript using the mean of the self-report scale. Scores range from 1-5 with higher scores indicating increased likeliness to miss doses of antiretroviral medication.
Time Frame: Day 1 post-test
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 64 | 66
score on a scale | 2.56 (1.43) | 2.53 (1.42)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Control | Intervention: 90 DAYS Film
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03898063/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT03898063/SAP_002.pdf
  • Informed Consent Form: Qualtrics Recruitment ICF (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03898063/ICF_003.pdf